CLINICAL TRIAL: NCT01369277
Title: A Phase 1, Randomized, Double Blind, Placebo-Controlled, Single Dose Escalation Study In Japanese Healthy Subjects, And Open Label, Single Dose Study In Western Healthy Subjects To Investigate The Safety, Tolerability, And Pharmacokinetics of PF-04991532.
Brief Title: A Single Dose Study In Japanese And Western Healthy Subjects To Investigate The Safety, Tolerability And Pharmacokinetics Of PF-04991532
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B2611013
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders
Keywords: PF-04991532; safety and tolerability; PK; Japanese and Western population
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders | interventions — 6-(3-cyclopentyl-2-(4-(trifluoromethyl)-1H-imidazol-1-yl)propanamido)nicotinic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Japanese cohort (Experimental): A total of 12 Japanese healthy subjects will be allocated to receive 3 ascending single doses (100 mg, 300 mg and 750 mg) of PF-04991532 or placebo through 3 dosing periods in a randomization ratio of 3:1.
  Interventions: Drug: PF-04991532; Drug: Placebo
- Weterner Cohort (Experimental): 9 western healthy subjects will be enrolled to receive 2 single ascending doses (300 mg and 750 mg) of PF-04991532 through 2 dosing periods.
  Interventions: Drug: PF-04991532

INTERVENTIONS:
Drug: PF-04991532 — Single dose administration of PF-04991532 (100 mg, 300 mg and 750 mg) in tablet formulation under fasted condition.
  Arms: Japanese cohort
Drug: Placebo — Single dose administration of matching placebo in tablet formulation at the fasted state
  Arms: Japanese cohort
Drug: PF-04991532 — Single dose administration of PF-04991532 (300 mg and 750 mg) in tablet formulation under fasted condition.
  Arms: Weterner Cohort

SUMMARY:
This study is to investigate the safety, tolerability and pharmacokinetics of single ascending oral doses of PF-04991532 in Japanese healthy subjects. The secondary objective is to investigate the pharmacokinetics and safety of single ascending oral doses of PF-04991532 in Western healthy subjects and to compare the pharmacokinetics between Japanese and Western healthy subjects.

DETAILED DESCRIPTION:
Safety/Tolerability and Pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential, between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight > 50 kg (110 lbs).
* Japanese subjects must have four Japanese grandparents who were born in Japan.
* Mean body weight and the body weight range of Western subjects must be within ±10% of the Japanese subjects.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Screening supine blood pressure >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), on a single measurement (confirmed by a single repeat, if necessary) following at least 5 minutes of rest.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
* Pregnant or nursing females or women of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10,12 and 16, 24, 36 and 48 hours post dose
Time for Cmax (Tmax) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10,12 and 16, 24, 36 and 48 hours
Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (AUClast) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10,12 and 16, 24, 36 and 48 hours
Area under the plasma concentration-time profile from time zero to 24 hours (AUC0-24) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10,12 and 16, 24, 36 and 48 hours
Total amount of unchanged drug excreted in the urine over 24 hours, expressed as percent of dose (Ae24%) | Urine collection from 0 to 24 hours post dose
Renal clearance (CLr) | Urine collection from 0 to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611013&StudyName=A%20Single%20Dose%20Study%20In%20Japanese%20And%20Western%20Healthy%20Subjects%20To%20Investigate%20The%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20PF-04991532